CLINICAL TRIAL: NCT03967704
Title: Optimization of Follow-up of Patients With Symptomatic Recent Osteoporotic Vertebral Fracture
Acronym: OPTIVERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPTIVERT
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Osteoporotic Fractures
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Life quality evaluation (Experimental): Patients consulting the Emergency Department (SAU) or the rheumatology department of the GHPSJ (referred by a colleague orthopaedic surgeon, rheumatologist, radiologist or other) for a recent symptomatic osteoporotic dorsal or lumbar vertebral fracture, are called for a rheumatology consultation, vertebral fracture consultation.
  Patients consulting in the rheumatology department during a spinal fracture consultation at the GHPSJ as well as patients hospitalized in the rheumatology department at the GHPSJ are selected consecutively.
  - Arm 1 (intervention): two additional consultations with the rheumatology
  Interventions: Procedure: Life quality evaluation

INTERVENTIONS:
Procedure: Life quality evaluation — As part of this research, 2 additional consultations at 12 months and 24 months will be carried out by one of the rheumatologists in the department. At the consultation 12 months after his inclusion, the patient will have a clinical examination, a quality of life questionnaire to complete and additional images (x-rays). For the 24-month consultation, the patient will have a clinical examination, a quality of life questionnaire to complete and the patient may have an additional X-ray of the spine if there is height loss > 2 cm and/or pain.

SUMMARY:
The management of osteoporotic fractures has recently changed with the emergence of new programs dedicated to the diagnosis and treatment of osteoporosis. For example, the Fracture Network of the Paris Saint-Joseph Hospital Group, created in 2015, identifies and ensures the care of patients who have consulted emergency rooms for osteoporotic fractures. Within this sector, the vertebral fracture (VF) appears to be the most frequent (22.4%) ahead of other fracture sites, confirming the results of other studies that consider VF as a real public health problem.

Osteoporotic vertebral fractures (OVF) have certain specificities compared to other osteoporotic fractures, encouraging particular interest.

DETAILED DESCRIPTION:
A. Particularities of OVF management

* Pain intensity caused by OVF justifies specific analgesic management. Analgesic management is sometimes complicated by co-morbidities and patients age, with poor analgesics tolerance, in particular opioids.
* OVF is responsible for a change in patients' quality of life, often with a loss of autonomy.
* VF is considered as severe fracture that warrants anti-osteoporotic drug therapy (if osteoporotic origin has been confirmed), in order to avoid risk of a new osteoporotic fracture.
* Progressive profil of pain associated with OVF and importance vertebral extent collapse may justify the use of specific "vertebral augmentation" procedures on vertebra, such as cementoplasty or kyphoplasty. These interventions are aimed at disappearance / reduction of pain related to OVF, improvement of life quality or correction or elimination of a static spinal disorder related to fracture.

B. Current rheumatology OVF management at the GHPSJ Patients management with OVF can be either outpatient or inpatient, depending on the extent of pain, fracture context, and co-morbidities.

- Rheumatology department of the GHPSJ has set up an outpatient patient path dedicated to osteoporotic vertebral fracture, making it possible to optimize patients concerned management. This route has follow characteristics : Patients with OVF are seen by rheumatologist during a consultation dedicated to OVF (Vertebral Fracture Consultation), and benefit the same day from spinal radiographs, bone densitometry and a biological assessment of fragile osteopathy on the GHPSJ site. During consultation, fracture history, risk factors for falls, bone history, an assessment of the patient's pain, functional abilities and life quality are performed. A spinal orthosis can be made if necessary.

Then patients are seen again 15 days later by the same rheumatologist with all results of the assessment During this 2nd consultation, depending on results of the additional examinations and patient's clinical progress, analgesic treatment is adapted. In addition, anti-osteoporotic treatment may be prescribed.

* For patients with OVF requiring hospital management in the rheumatology department, additional examinations are also carried out with the same anamnestic and clinical elements as for the above-mentioned outpatient management. Nevertheless, intensity of pain may initially prevent certain additional examinations, such as bone densitometry, from being carried out, which in this case are deferred until the patient's state of health allows them.
* During outpatient or inpatient journey, depending on results of additional examinations and patient's clinical progress, intervention therapy can be decided and carried out as soon as possible (cementoplasty). Patients for whom cementoplasty is performed are hyperalgia patients with rapid loss of autonomy due to vertebral fracture and a general condition compatible with general anesthesia. Following cementoplasty, patients are seen again in consultation for 1 month for a clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Patient consulting or hospitalized in the rheumatology department at the GHPSJ for recent and symptomatic osteoporotic spinal or lumbar fracture Recentness is defined either by anamnestic event existence (example: fall) to date the fracture less than 4 months old, or by MRI or CT signs existence of attesting to recent nature of the fracture: hypersignal T2 stir & hyposignal T1 on MRI, presence of a cleft on the CT, on imaging less than 4 months old.

Symptomatic is defined as spinal pain existence in relation to the vertebral fracture, not attributable to any cause other than the fracture.

* Patient affiliated to a health insurance plan
* Patient capable of giving free, informed and express consent

Exclusion Criteria:

* Patient with fractures occurring on metastatic spine
* Patient with unstable VF, requiring rapid orthopedic management
* Patient with a history of cementoplasty on dorsal or lumbar spine
* Patients transferred to another hospital after transition to SAU
* Homeless patient
* Patient not residing in Ile-de-France
* Patient who is bedridden or has one or more severe co-morbidity(s) that puts fractured osteoporosis in background
* Patient deprived of liberty
* Patient under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Assess life quality of patients with osteoporotic VF 12 months after symptomatic vertebral fracture diagnosis: Quality of life questionnaires (QUALEFFO-41) | 1 year
  Quality of life questionnaires (QUALEFFO-41)

SECONDARY OUTCOMES:
Assess pain related to vertebral fracture at D0, M12 and M24 after diagnosis: Analogical visual scale | Day 0 - 1 year - 2 years
  Analogical visual scale on the pain and taking painkillers (yes/no)
Assess life quality: Quality of life questionnaires (QUALEFFO-41) | 2 years
  Quality of life questionnaires (QUALEFFO-41)
Measurement of the walking perimeter | Day 0 - 1 year - 2 years
  the maximum distance that the person can travel without stopping (in meters)
Number of new osteoporotic fractures (vertebral or nonvertebral) | 1 year - 2 years
  Fractures that have been confirmed by an imaging examination (X-ray, +- MRI or CT)
Number of new fall(s) | 1 year - 2 years
Number of hospitalizations for all causes | 1 year - 2 years
Spinal statics | 1 year - 2 years
  Height in centimeters
Management of osteoporosis | 1 year - 2 years
  prescription completed (yes/no) antiosteoporotic treatment taken (yes/no)
Analogical visual scale of patient satisfaction | 1 year - 2 years
  (scale of 0 to 10) following the information meeting with a nurse on osteoporosis

CONTACTS AND LOCATIONS:
Overall Officials: Agnès PORTIER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Ballane G, Cauley JA, Luckey MM, El-Hajj Fuleihan G. Worldwide prevalence and incidence of osteoporotic vertebral fractures. Osteoporos Int. 2017 May;28(5):1531-1542. doi: 10.1007/s00198-017-3909-3. Epub 2017 Feb 6. PMID 28168409
- [Result] Venmans A, Lohle PN, van Rooij WJ. Pain course in conservatively treated patients with back pain and a VCF on the spine radiograph (VERTOS III). Skeletal Radiol. 2014 Jan;43(1):13-8. doi: 10.1007/s00256-013-1729-x. Epub 2013 Oct 8. PMID 24100705
- [Result] Jung HJ, Park YS, Seo HY, Lee JC, An KC, Kim JH, Shin BJ, Kang TW, Park SY. Quality of Life in Patients with Osteoporotic Vertebral Compression Fractures. J Bone Metab. 2017 Aug;24(3):187-196. doi: 10.11005/jbm.2017.24.3.187. Epub 2017 Aug 31. PMID 28955695
- [Result] Lips P, Cooper C, Agnusdei D, Caulin F, Egger P, Johnell O, Kanis JA, Liberman U, Minne H, Reeve J, Reginster JY, de Vernejoul MC, Wiklund I. Quality of life as outcome in the treatment of osteoporosis: the development of a questionnaire for quality of life by the European Foundation for Osteoporosis. Osteoporos Int. 1997;7(1):36-8. doi: 10.1007/BF01623457. PMID 9102060
- [Result] Lindsay R, Silverman SL, Cooper C, Hanley DA, Barton I, Broy SB, Licata A, Benhamou L, Geusens P, Flowers K, Stracke H, Seeman E. Risk of new vertebral fracture in the year following a fracture. JAMA. 2001 Jan 17;285(3):320-3. doi: 10.1001/jama.285.3.320. PMID 11176842
- [Result] Li L, Ren J, Liu J, Wang H, Wang X, Liu Z, Sun T. Results of Vertebral Augmentation Treatment for Patients of Painful Osteoporotic Vertebral Compression Fractures: A Meta-Analysis of Eight Randomized Controlled Trials. PLoS One. 2015 Sep 17;10(9):e0138126. doi: 10.1371/journal.pone.0138126. eCollection 2015. PMID 26378444
- [Result] Carlier RY, Gordji H, Mompoint DM, Vernhet N, Feydy A, Vallee C. Osteoporotic vertebral collapse: percutaneous vertebroplasty and local kyphosis correction. Radiology. 2004 Dec;233(3):891-8. doi: 10.1148/radiol.2333030400. Epub 2004 Oct 14. PMID 15486209
- [Result] Tsoumakidou G, Too CW, Koch G, Caudrelier J, Cazzato RL, Garnon J, Gangi A. CIRSE Guidelines on Percutaneous Vertebral Augmentation. Cardiovasc Intervent Radiol. 2017 Mar;40(3):331-342. doi: 10.1007/s00270-017-1574-8. Epub 2017 Jan 19. PMID 28105496
- [Result] Ibrahim A, Singh DKA, Shahar S. 'Timed Up and Go' test: Age, gender and cognitive impairment stratified normative values of older adults. PLoS One. 2017 Oct 3;12(10):e0185641. doi: 10.1371/journal.pone.0185641. eCollection 2017. PMID 28972994
- [Result] Genant HK, Wu CY, van Kuijk C, Nevitt MC. Vertebral fracture assessment using a semiquantitative technique. J Bone Miner Res. 1993 Sep;8(9):1137-48. doi: 10.1002/jbmr.5650080915. PMID 8237484